CLINICAL TRIAL: NCT02235220
Title: Reduction of Masticatory Muscle Activity by Restoring Canine Guidance With Composite Resin Fillings in Patients With Bruxism.
Brief Title: Reduction of Masticatory Muscle Activity by Restoring Canine Guidance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Martin Sasse, Dr. Martin Sasse, D.M.D, Assistant Professor, University of Kiel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Canine guidance / Grindcare; D 432/12 (Other: Ethics Commission University of Kiel, Germany)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Bruxism; Myopathy; Muscular Activity
Keywords: Bruxism
MeSH Terms: conditions — Bruxism; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Composite resin restoration (Experimental): A canine guidance is reestablished by additive composite resin restorations of the canine cusp.
  Interventions: Other: Composite resin restoration

INTERVENTIONS:
Other: Composite resin restoration — Masticatory muscular activity is measured before and after treatment with additive composite resin fillings (Tetric EvoCeram, Ivoclar Vivadent, Schaan, Liechtenstein). A Grindcare (Medotech A/S, Herlev, Denmark) device is used for determination of muscular activity.
  A first measurement is conducted, followed by 4 weeks without any intervention. A second measurement is then carried out before restoration of the canine cusps with composite fillings. A third measurement is conducted, again followed by 4 weeks without any intervention. At last a final measurement is conducted.

SUMMARY:
In this study it is to be evaluated wether a restoration with composite resin fillings to reestablish a canine guidance will reduce masticatory muscle activity in patients with bruxism.

DETAILED DESCRIPTION:
30 patients showing clinical symptoms of bruxism receive treatment within this clinical trial. Typical symptoms like pain or tenseness of the masticatory muscles, headache or abrasions are mandatory preconditions. Exclusion criteria are a present treatment with a biteguard or a sufficient canine guidance.

In the first session a detailed history, a dental status and a clinical functional status are recorded. The baseline situation is documented by taking impressions with alginate of the maxilla and mandible for diagnostic study models. Following this procedure a first measurement of the muscular activity is conducted for seven days with the Grindcare device.

After four weeks without any intervention a second measurement is conducted again for seven days.

In the next session the canine cusps are restored with composite fillings. Finally a sufficient canine guidance should be present. In the same session a second impression of the maxilla is taken. A third measurement is conducted, again followed by four weeks without any intervention.

At last another impression of the maxilla is obtained and a final measurement for seven days is conducted.

At the first examination and after the third measurement of the masticatory muscle activity the patients fill out the questionnaire of the Oral Health Impact Profile in order to allow for the assessment of possible functional restraints and mental interferences.

ELIGIBILITY:
Inclusion Criteria:

* patients show signs of bruxism
* no canine guidance is present
* no prosthodontic restorations of the canine are present

Exclusion Criteria:

* a sufficient canine guidance is present

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of masticatory muscular activity | 13 weeks
  Masticatory muscular activity is measured before and after treatment with additive composite resin fillings (Tetric EvoCeram, Ivoclar Vivadent, Schaan, Liechtenstein). A Grindcare (Medotech A/S, Herlev, Denmark) device is used for determination of muscular activity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kern, DDS, PhD, Study Director — University of Kiel